CLINICAL TRIAL: NCT05976958
Title: Utility and Validation's Study of a Smartphone Application for Periodic Paralysis
Acronym: RaDiCo-PP
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C16-99; 2017-A01827-46 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2023-07-18; First posted 2023-08-04 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Periodic Paralyses
Keywords: Periodic paralyses; Quality of life; Rare disease
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Periodic paralyses (PP) are rare genetic disorders characterized by the occurrence of acute and reversible episodes of muscle weakness. Their episodic and highly variable nature makes it difficult to gather the necessary information for monitoring and therapeutic adaptation. Patients struggle to accurately report the number, duration, severity, and triggers of their attacks that have occurred between two consultations.

Currently, there are no validated scales or tools for precisely and standardizedly assessing paralytic episodes. Ecological Momentary Assessment (EMA) is a real-time data collection method used in research, historically on paper forms and then on expensive and cumbersome electronic devices (PDAs). The widespread use of smartphones opens up a new avenue in this field, and the use of a mobile application as a real-time data collection tool could be perfectly applicable to these conditions with episodic expression. It is hypothesized that systematic and real-time collection of paralysis episode characteristics will improve the quality and accuracy of the collected data, thus enhancing clinicians' understanding of the condition and patient management. Moreover, little is known about the medical and social impact of the disease. To address these specific issues, the investigators propose a study of patients with "Periodic Paralyses" based on prospective collection of clinical and medico-social data during routine consultations and in real-time during paralytic episodes using a dedicated smartphone application developed by Ad Scientiam in collaboration with Dr. Savine Vicart, the study coordinator.

The primary objective of this study is to evaluate the benefit of a smartphone application specifically developed for patients with periodic paralyses to collect real-time information and improve the quality of collected data regarding the characteristics of paralysis episodes (number, duration, intensity, triggering factors, location, treatment) compared to the retrospective questionnaire typically used in consultations.

The secondary objective is to assess the impact of this new data collection method on the medical management of patients.

DETAILED DESCRIPTION:
Primary periodic paralyses (PP) are rare autosomal dominant disease (estimated prevalence of one per 100.000 in Europe) due to mutations in genes encoding muscle ion channels. Symptoms usually start in childhood or adolescence. They are characterized by acute and reversible muscle weakness attacks. The features of paralytic attacks (severity, frequency, duration, triggering factors) are highly variable. Thus, for a given patient, the weakness can:

Be focal (involving only one limb) or generalized (para or tetraplegia) with sometimes some swallowing and breathing difficulties; Last minutes / hours to several days; Occur very episodically (e.g. several months apart) and then daily and be spaced again; Be triggered by immobility, rest after strenuous exercise, dietary factors, cold, stress, infections, hormonal variations, specific medications like corticosteroids.

However, exposure to these risk factors does not systematically trigger a crisis.

After an initial phase dominated by attacks of transient flaccid paralysis, a persistent and progressive weakness may occur, in addition to the attacks of weakness, that is related to a limb-girdle vacuolar myopathy . It is unclear whether this is directly related to the frequency and severity of the episodes of weakness.

Classically, PP are classified as hyperkalemic (hyperPP) or hypokalemic (hypoPP) based on changes in blood potassium levels during the access. These changes are often subtle and transient making the distinction between the 2 forms difficult. If this serum potassium-based classification is clinically useful, it is not correlated to the genes identified to be responsible of PP. Thus, mutations in different genes can lead to a same phenotype and different mutations in a same gene lead to distinct phenotypes.

3 genes (CACN1AS, SCN4A and KCNJ2) have been identified in PP HypoPP is the most common PP. Inheritance is autosomal dominant with reduced penetrance in woman. Symptoms typically begin in the second decade. Attacks of paralysis usually occur on awakening in the night or in the early morning, last for hours (occasionally days) with gradual resolution and are provoked more specifically by rest after exercise and carbohydrate-rich meals. Mutations in the alpha subunit of the skeletal muscle calcium channel gene CACN1AS cause most cases (70%). Approximatively, 10-20% are due to mutations in the voltage-gated sodium channel gene SCN4A. So, a small number of affected individuals do not have a mutation in these 2 genes and are not linked to these loci. HyperPP is due to mutations in SCN4A encoding the alpha subunit of the skeletal muscle voltage- gated sodium channel. Onset of episodic weakness is commonly observed earlier than for HypoPP (first decade). In contrast with HypoPP, the attacks frequently occur during the daytime but nocturnal access may happen, last few minutes to hours and are mostly triggered by cold, rest after exercise and fasting. Electrical myotonia is found in 50% off affected individuals but is clinically apparent in less than 20%.

Andersen-Tawil Syndrome (ATS) is characterized by the triad, often incomplete, of PP (hypo or hyperPP), ventricular arrhythmia and distinctive physical features. It is the least common form of PP. Mutations in KCNJ2 encoding the inward rectifying potassium channel kir2.1 have been identified in about two-thirds of patients with ATS.

The development of functional electromyographic (EMG) tests has revolutionized the diagnostic approach for channelopathies in general and for PP in particular. These tests are based on an EMG examination that measures the amount of muscle's actions potentials (CMAPs) under conditions that reproduce the conditions of induction of paralytic attacks (brief repeated exercises, long exercise, cooling test). It shows two distinct patterns predictive of mutations found by the molecular diagnosis in 85% of cases. It is now good practice to perform a functional EMG prior to molecular diagnosis. The combination of EMG and molecular diagnosis allows an effective diagnosis of periodic paralysis.

Treatment mostly relies on advices such as avoiding triggering factors or dietary recommendations. Potassium chloride can be used for acute attack in hypoPP and regular use may reduce its frequency. Inhibitors of carbonic acid anhydrase (acetazolamide, dichlorphenamide) are usually helpful in all forms of PP.

Thereby, diagnosis, monitoring and management of PP are complex. This justified the labellisation of our team in 2005 in National Channelopathies Reference Center. The investigators work at national level in collaboration with the other French Neuromuscular Centres from the "filière neuromusculaire" and coordinate the national network on channelopathies named RESOCANAUX. The investigators collaborate with the international teams from North America (USA, Canada) and Europe (Italy, Netherlands, England) grouped within the Muscle Society Group (MSG) coordinated by Prof. Griggs, Rochester, USA.

Our experience with patients and their families led us to the following observations:

The collection of information necessary for the patient's follow-up and for therapeutic adjustments is complicated by the episodic and highly variable expression of the symptoms. At each follow-up visits, patients struggle to accurately report the number, duration, severity and triggering factors of their crises which have occurred within the range of 2 out-patient visits. Currently, the usual tool of data communication between patients and clinicians is, at best, patient's paper diary. It is often perceived as a boring document and therefore fill in compliance is poor. Retrospective or generalized responses are, to a significant degree, inaccurate because of limitations in autobiographical memory whereby respondents must rely on estimation, extrapolation and inference strategies that are inherently unreliable. Thereby, in such cases, patients under-report their attacks and clinicians have limited information to recommend the appropriate treatment.

The difficulties of locomotion resulting from paralysis and their repetition over time lead to social and economic consequences, such as : (1) a frequent professional or school absenteeism leading to grade repetitions, establishment of remedial classes..; (2) organization of catch-up sessions for exams in case of absenteeism to the regular session; (3) difficulties to deal with job involving physical activity or out-door exposure (weather effect) leading to job eviction or professional relocation ; (4) a more complex choice for the socio- professional sector ...

During paralytic attacks, patients are dependent on someone for several hours for most activities of daily life (movements, hygiene, and elimination, feeding...). This impacts strongly caregivers' life (spouses, parents or other ...) even more if there are several patients in the same household. Thus, caregivers stay at home to take care for their children /spouses and their absenteeism adds to the patients' ones.

Thus, it appears crucial to succeed in assessing more accurately both the clinical and medico- economic impacts of these pathologies to improve, in the future, healthcare and healthcare costs.

Currently, there is no validated scale or tool to assess paralytic attacks in a precise and standardized way. Ecological momentary assessment (EMA) refers to a collection of methods often used in medicine research by which a participant repeatedly reports on symptoms close in time to experience and in the participants' natural environment. This collection method has historically been under-utilized as it was performed on imprecise paper-logs that patients filled at home. For the last 10-15 years EMA studies migrated to electronic medias (PDAs) but these (1) require participants to become familiar with and carry a device they would otherwise not carry, (2) remain expensive and hard to implement on large-scale studies, (3) require programming expertise and (4) oblige to provide a device to each participant. The generalization of the Smartphone in the population opens a new avenue of research in the field of EMA because of: (1) their lower cost, (2) the widespread adoption of phones with increasingly powerful technical capabilities (de facto pocket computers), (3) people's tendency to carry their phones everywhere, (4) people's attachment to their phones and (5) context awareness features enabled through sensing and phone-based personnel information. In 2013, there were 27 million of smartphone owners in France which corresponds to 50% of the French population aged 11 and over, according to the quarterly barometer made by the Mobile Marketing Association France, in partnership with comScore, GFK and Médiamétrie. In 2014, it was sold twice more tablets than laptops (7.9 million against 3.7) and more than 17 million Smartphones.

The use of a mobile application as a tool for real-time data collection could fit perfectly to the pathologies with episodic expression like periodic paralysis and holds promise for making self- assessment/monitoring easier.

The investigators hypothesize that systematic and prospective data collection of the features of periodic paralytic attacks through a mobile application will improve the quality and precision of the collected data, and therefore both clinicians and patients' knowledge of the disease and will consequently upgrade the current care of patients.

In addition, the investigators do not know much about the medico-social and economic impact of the disease.

To better tackle these specific issues, the investigators propose study of the population "Periodic Paralysis" followed in the National Channelopathies Reference Center based on a prospective collection of clinical and medico-economic data during follow-up visits scheduled as part of their usual care and in real-time via an EMA smartphone application.

ELIGIBILITY:
Inclusion Criteria:

All patients with periodic paralysis aged over 12 years and followed in the National Channelopathies Reference Centre will be eligible for the study if they:

are able to understand, read and write French

are willing to and capable of entering their clinical and medico-social and economic data in the Smartphone application

have an identified parent/caregiver for children aged 12-18 years (not mandatory for adults)

are affiliated to a Health Insurance

are able to give their informed consent (adult patients) or if their legal representatives are able to give their informed consent (child patients)

Exclusion Criteria: Will not be eligible, patients

with a condition that could explain hypokalemia: renal, adrenal, thyroid dysfunction, renal tubular acidosis, abuse of diuretic and laxative,

with a condition that could explain hyperkalemia: renal, adrenal, thyroid dysfunction, use of potassium-sparing diuretics,

who are under guardianship

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients over 12 years of age with periodic paralyses, being followed at the Muscular Channelopathies Reference Center at the Pitié-Salpêtrière Hospital Group, who meet the inclusion criteria, are adequately informed, and have provided consent, may be enrolled in the study by their physician.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Assessing the benefit of in-real-time data capture on quality of the collected informations, via a smartphone application, compared to retrospective collection via an interview during routine patient care visits | Through study completion, at 6 months, 12 months, and 18 months.
  The primary objective is to measure, for characteristics of paralysis attacks (number, duration, intensity, triggering factors, location, treatment), the benefit of in-real-time data capture on quality of the collected informations, via a smartphone application, compared to retrospective collection via an interview during routine patient care visits

SECONDARY OUTCOMES:
Assessing the benefit of in-real-time data capture on the characteristics of paralysis attacks (number, duration, severity) via a smartphone application, compared to retrospective collection via an interview during routine patient care visits. | Through study completion, at 6 months, 12 months, and 18 months.
  The secondary objective is to measure, for periodic paralysis patient care management, the benefit of in-real-time data capture on the characteristics of paralysis attacks (number, duration, severity) via a smartphone application, compared to retrospective collection via an interview during routine patient care visits.

CONTACTS AND LOCATIONS:
Overall Officials: Savine Vicart, Principal Investigator — INSERM U1127 - IHU- ICM
Locations (1):
- RaDiCo-PP, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided